CLINICAL TRIAL: NCT01856933
Title: BrUOG 263: PSMA ADC for Recurrent Glioblastoma Multiforme (GBM): A Phase II Brown University Oncology Research Group Study
Brief Title: BrUOG 263: Prostate Specific Membrane Antigen (PSMA) Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich Elinzano, MD (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry); Rhode Island Hospital (Other); University of Texas (Other)
Responsible Party: Sponsor-Investigator, Heinrich Elinzano, MD, Prinicipal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 263
Record Dates: First submitted 2013-01-08; First posted 2013-05-20 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: GBM; Glioblastoma Multiforme; Gliosarcoma
Keywords: GBM; Glioblastoma Multiforme; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — PSMA ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PSMA ADC (Experimental): 2.5 mg/kg, IV, over 60 minutes every 3 weeks
  Interventions: Drug: PSMA ADC

INTERVENTIONS:
Drug: PSMA ADC — 2.5 mg/kg, IV, over 60 minutes every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Prostate Specific Membrane Antigen (PSMA ADC), as well as its safety and side effects for patients with advanced brain tumors. This study will also study how your body metabolizes (breaks down) PSMA ADC.

DETAILED DESCRIPTION:
PSMA expression has been demonstrated in the tumor neovasculature of Glioblastoma Multiforme (GBM) by immunohistochemical staining. Strong reactivity to the antibody component of PSMA ADC was observed in the endothelial cells of new tumor blood vessels in GBM. Since the endothelial cells are located on the luminal surface of blood vessels, PSMA ADC does not need to cross the blood brain barrier to reach its target. Following binding and internalization of PSMA ADC, the cytotoxic component of PSMA ADC will be released and destroy the neovasculature that supports tumor growth. Therefore, PSMA ADC may be an active treatment for GBM.

Bevacizumab, an inhibitor of angiogenesis, has been shown to be effective in improving progression-free survival as a single agent. Thus PSMA ADC, which targets tumor angiogenesis by a mechanism different from that of bevacizumab, may be a novel therapeutic modality for GBM.

A phase 2 study of PSMA ADC is proposed for patients with GBM that have progressed after standard treatment that includes radiation, temozolomide and bevacizumab. A phase 1 study of PSMA ADC in prostate cancer is ongoing and a phase 2 dose level of 2.5 mg/kg IV every 3 weeks has been defined. Treatment after bevacizumab failure for patients with GBM is a major unmet medical need. If activity were demonstrated in this trial, a definitive randomized study would be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Males and females Histologically confirmed GBM (Patients with gliosarcoma are also eligible)
* Assessable or measurable disease by MRI
* Progression after prior treatment that includes radiation, temozolomide and bevacizumab.

  -> 4 weeks since prior chemotherapy, bevacizumab and other systemic treatment and > 3 weeks from prior radiation.
* age >18 years
* Weight < 150 kg.
* Karnofsky performance score > 60
* Life expectancy >12 weeks
* Brain MRI within 21 days prior to registration
* Laboratory results requirements

  * Absolute neutrophil count (ANC) ≥ 1000/mm3.
  * Platelets (Plt) ≥ 100,000/mm3
  * Hemoglobin (Hgb) ≥ 8.0 g/dL
  * Total bilirubin ≤ 2.0 mg/dL
  * Serum alanine transferase/ Serum aspartate transaminase (ALT/AST) ≤ 2.5x the upper limit of normal (ULN)
  * Serum creatinine ≤ 2.0 mg/dL
  * Pancreatic Amylase (p-amylase) ≤ the ULN
  * Negative serum pregnancy test for women of child-bearing potential
* Stable corticosteroid dose at least 14 days prior to registration
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients must not be on enzyme-inducing anti-epileptic drugs (EIAED). Patients may be on non-enzyme inducing anti-epileptic drugs (NEIAED) or may not be taking any anti-epileptic drugs. A list of AED that cause modest or no induction of hepatic metabolic enzymes will be discussed

Exclusion Criteria:

* Non-GBM primary invasive malignant neoplasm within the five years prior to screening except for:

  * keratinocyte (non-melanoma) (i.e., basal cell, squamous cell) carcinoma of the skin; or low-grade papillary superficial transitional cell carcinoma of the bladder.However, patients with stage 1 cancers not requiring cancer therapy including chemotherapy or hormone therapy, for which a lifespan of greater than 3 years without treatment is expected (such as early stage prostate cancer) may be enrolled.
* Clinically significant cardiac disease (New York Heart Association Class III/ IV or severe debilitating pulmonary disease
* Subjects with QTc>500 msec (either Bazzett's or Fridericia's method)
* Radiation therapy, cytotoxic chemotherapy, bevacizumab or other treatment for GBM within previous three weeks
* Evidence of an active infection requiring ongoing intravenous antibiotic therapy
* Any toxicity ≥ grade 2 (non-laboratory) (NCI CTCAE, Version 4.03) prior to first dose of study drug
* Prior treatment with PSMA ADC or other therapies targeting PSMA, or other anti-body drug conjugate (ADC) products that contain monomethyl auristatin E (MMAE) (e.g., brentuximab vedotin, glembatumumab vedotin, ASG-5ME)
* Known hypersensitivity reactions to PSMA ADC or any of its components.
* Any medical condition that in the opinion of the Investigator may interfere with a subject's participation in or compliance with the study
* Patients with a prior history of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Elinzano, MD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Southwestern, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PSMA ADC
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PSMA ADC
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [39 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Progression) for Patients With Glioblastoma That Have Progressed After Prior Treatment That Has Included Radiation, Temozolomide and Bevacizumab.
Description: The response assessment in neuro-oncology (RANO) will be used to define radiographic response.
  (PD): A >25% increase in tumor area (product of two diameters) OR appearance of a new lesion/site, OR clear clinical worsening or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 3 months until progression, potentially up to 1 year
Population: Progression
Measure: Number; unit: participants
Arm/Group | PSMA ADC
Number analyzed (Participants) | 6
participants | 6

2. Secondary Outcome: Number of Patients Who Experienced Toxicities (Adverse Events) Who Received PSMA ADC for Recurrent Glioblastoma.
Description: Please note that toxicities outlined may not all be related to the treatment regimen.
Time Frame: at least every 3 weeks for a maximum of 30 post coming off drug, approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | PSMA ADC
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Arm/Group | PSMA ADC
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSMA ADC (N=6)
eye disorder/ vision changes (Investigations) | 1 (1)
H/A (Investigations) | 1 (1)
Hypermagnesemia (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Intratumoral hemorrhage (Investigations) | 1 (1)
Nausea (Investigations) | 1 (1)
Thrombocytopenia (Investigations) | 2 (2)
seizure (Investigations) | 1 (1)
UTI (Investigations) | 1 (1)
WBC (Investigations) | 1 (1)
confusion (Investigations) | 1 (1)
muscle weakness/weakness general (Investigations) | 2 (2)
dyspnea (Investigations) | 1 (1)
Facial muscle weakness (Investigations) | 1 (1)
CD4 Lymph count (Investigations) | 2 (2)
Lymphopenia (Investigations) | 1 (1)
Anorexia (Investigations) | 1 (1)
syncope (Investigations) | 2 (2)
pain (Investigations) | 1 (1)
perforation-sigmoid (Investigations) | 1 (1)
cholesterol (Investigations) | 1 (1)
creatinine (Investigations) | 1 (1)
hyperglycemia (Investigations) | 1 (1)
hypoalbumin (Investigations) | 1 (1)
troponin (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSMA ADC (N=6)
AKI (Investigations) | 1 (1)
Alopecia (Investigations) | 1 (1)
ALT (Investigations) | 2 (2)
AST (Investigations) | 1 (1)
anemia (Investigations) | 1 (1)
edema, lower leg (Investigations) | 1 (1)
eye disorder/ vision changes (Investigations) | 1 (1)
fatigue (Investigations) | 2 (2)
H/A (Investigations) | 1 (1)
Hypermagnesemia (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Hyponatremia (Investigations) | 2 (2)
Infection/shingles/thrush (Investigations) | 2 (2)
Nausea (Investigations) | 1 (1)
Neutrophil count (Investigations) | 1 (1)
Thrombocytopenia (Investigations) | 2 (2)
vomiting (Investigations) | 1 (1)
rash- torso (Investigations) | 1 (1)
parathesia/neuropathy (Investigations) | 1 (1)
rash- papular (Investigations) | 1 (1)
urinary incontinence (Investigations) | 1 (1)
right ankle swelling (Investigations) | 1 (1)
UTI (Investigations) | 1 (1)
WBC (Investigations) | 3 (3)
intracerebral hematoma (Investigations) | 1 (1)
Lymphopenia (Investigations) | 2 (2)
dysphasia (Investigations) | 2 (2)
gait disturbance (Investigations) | 1 (1)
cognitive disturbance/impairment (Investigations) | 2 (2)
dysgeusia (taste) (Investigations) | 1 (1)
pain- left calf/leg (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No